CLINICAL TRIAL: NCT02268032
Title: Assess the Effect of DHEA or Other Androgenic Agents on Ovarian Reserve Markers in Women With Diminished Ovarian Reserve
Brief Title: Assess the Effect of Dehydroepiandrosterone (DHEA) or Other Androgenic Agents Over Markers of Ovarian Reserve
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DVR+T001
Record Dates: First submitted 2014-08-25; First posted 2014-10-20 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Healthy Women; Infertility, Female
Keywords: Hormone replacement therapy
MeSH Terms: conditions — Infertility, Female | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaginal ring 1 (VRD) (Experimental): 20 women using DHEA (VRD) for 2 menstrual cycles
  Interventions: Drug: DHEA
- Vaginal ring 2 (VRaA) (Experimental): 20 women using another androgenic agent (VRaA) for 2 menstrual cycles
  Interventions: Drug: Another Androgenic Agent (VRaA)
- Vaginal ring 3 (VR2A) (Experimental): 20 women using fixed combination of 2 androgenic agents (VR2A) for 2 menstrual cycles
  Interventions: Drug: Fixed combination of 2 androgenic agents (VR2A)

INTERVENTIONS:
Drug: DHEA — DHEA 2.2 g in vaginal ring
  Arms: Vaginal ring 1 (VRD)
Drug: Another Androgenic Agent (VRaA) — Testosterone 35 mg in vaginal ring
  Arms: Vaginal ring 2 (VRaA)
Drug: Fixed combination of 2 androgenic agents (VR2A) — DHEA 1.5 g/testosterone 25 mg fixed combination in vaginal ring
  Arms: Vaginal ring 3 (VR2A)

SUMMARY:
This study was conducted to evaluate the effect of a continuous administration of dehydroepiandrosterone (DHEA) or other androgenic agents on ovarian reserve markers in women with diminished ovarian reserve (ROD), such as antral follicle count (AFC) and anti-Müllerian hormone (AMH) concentrations.

DETAILED DESCRIPTION:
Healthy women attending the clinic of the Mother and Health Research Institute (IDIMI) were invited to participate, if they could not become pregnant due to surgical sterilization, and if they presented no contraindications to use androgen therapy.

Project Objectives :

The general objective was to evaluate pharmacokinetic parameters of three vaginal rings containing DHEA, testosterone, or combination of both hormones in women.

Secondary objectives were to assess effects on the hormonal profile, tolerability and incidence of adverse events.

* DHEA and/or, testosterone levels
* Estradiol, follicle stimulating hormone (FSH), sex hormone binding globulin (SHBG), androstenedione, morning cortisol, insulin growth factor 1 (IGF-1) levels
* Tolerability and safety assessment by the use of the vaginal ring.
* The incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Women between 38 and 45 years of age who have not used hormonal contraceptive methods at least for the past two months, or who have been surgically sterilized, with no contraindications for androgenic therapy.
2. Women with preserved menstrual cycles.
3. Women smoking less than 5 cigarettes daily.
4. Anti-Müllerian hormone (AMH) between 0.5-1.1 ng/mL
5. Total antral follicle count (AFC) 5-7

Exclusion Criteria:

1. Women receiving medications that interact with DHEA metabolism (Anastrozole, exemestane, Fulvestrant, Insulin, Letrozole, Tamoxifen, Triazolam).
2. Women with diabetes mellitus
3. Women with untreated or decompensated endocrine disorders
4. Women with a prior history of ovarian surgery or oophorectomy

Ages: 38 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of the association of DHEA plus testosterone over ovarian reserve markers | Before therapy start and up to 2 months thereafter
  The ovarian reserve markers antral follicle count (AFC) and anti-Müllerian hormone (AMH) were determined before and after hormonal therapy to compare the levels of both hormones between mono- and combination therapy and to investigate a potentially synergistic effect of the association of DHEA plus testosterone.

SECONDARY OUTCOMES:
Plasma levels of sex hormone binding globulin (SHBG), androstenedione, morning cortisol, insulin growth factor 1 (IGF-1), testosterone, dehydroepiandrosterone, follicle stimulating hormone (FSH), and estradiol | Before therapy start and up to 2 months thereafter
  A composite of hormones was measured and compared before and after hormonal therapy.
Tolerability of using the vaginal ring | After therapy start (vaginal ring insertion) and after 2 months (ring extraction)
  A questionnaire was used post insertion and post extraction of the vaginal ring to assess tolerability. The following was addressed: changes in vaginal discharge (never happened/no change/increased a little/increased much/changed color), vaginal infection (by fungi or bacteria: yes/no), burning (yes/no), odor (yes/no), pain (yes/no; if yes, assessed on a 1 to 10 scale for no pain to worst pain), discomfort (yes/no) or dryness (yes/no) of the vagina, changes (for couples) in the sexual relationship by the use of the vaginal ring (better/as always/with annoyance/with pain/did not have).
Number of subjects with adverse events per treatment group | From therapy start to up to 2 months
  Adverse events were collected by non-leading questions.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Mother and Health Research Institute (IDIMI), Faculty of Medicine, University of Chile, Santiago, International, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander JL, Kotz K, Dennerstein L, Kutner SJ, Wallen K, Notelovitz M. The effects of postmenopausal hormone therapies on female sexual functioning: a review of double-blind, randomized controlled trials. Menopause. 2004 Nov-Dec;11(6 Pt 2):749-65. doi: 10.1097/01.gme.0000142887.31811.97. PMID 15543027
- [Background] Barad D, Gleicher N. Effect of dehydroepiandrosterone on oocyte and embryo yields, embryo grade and cell number in IVF. Hum Reprod. 2006 Nov;21(11):2845-9. doi: 10.1093/humrep/del254. Epub 2006 Sep 22. PMID 16997936
- [Background] Balasch J, Fabregues F, Penarrubia J, Carmona F, Casamitjana R, Creus M, Manau D, Casals G, Vanrell JA. Pretreatment with transdermal testosterone may improve ovarian response to gonadotrophins in poor-responder IVF patients with normal basal concentrations of FSH. Hum Reprod. 2006 Jul;21(7):1884-93. doi: 10.1093/humrep/del052. Epub 2006 Mar 3. PMID 16517559
- [Background] Broekmans FJ, Soules MR, Fauser BC. Ovarian aging: mechanisms and clinical consequences. Endocr Rev. 2009 Aug;30(5):465-93. doi: 10.1210/er.2009-0006. Epub 2009 Jul 9. PMID 19589949
- [Background] Fabregues F, Penarrubia J, Creus M, Manau D, Casals G, Carmona F, Balasch J. Transdermal testosterone may improve ovarian response to gonadotrophins in low-responder IVF patients: a randomized, clinical trial. Hum Reprod. 2009 Feb;24(2):349-59. doi: 10.1093/humrep/den428. Epub 2008 Dec 3. PMID 19054777
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Gleicher N, Weghofer A, Barad DH. Improvement in diminished ovarian reserve after dehydroepiandrosterone supplementation. Reprod Biomed Online. 2010 Sep;21(3):360-5. doi: 10.1016/j.rbmo.2010.04.006. Epub 2010 Apr 18. PMID 20638339
- [Background] Pandian Z, McTavish AR, Aucott L, Hamilton MP, Bhattacharya S. Interventions for 'poor responders' to controlled ovarian hyper stimulation (COH) in in-vitro fertilisation (IVF). Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004379. doi: 10.1002/14651858.CD004379.pub3. PMID 20091563
- [Background] Wiser A, Gonen O, Ghetler Y, Shavit T, Berkovitz A, Shulman A. Addition of dehydroepiandrosterone (DHEA) for poor-responder patients before and during IVF treatment improves the pregnancy rate: a randomized prospective study. Hum Reprod. 2010 Oct;25(10):2496-500. doi: 10.1093/humrep/deq220. Epub 2010 Aug 21. PMID 20729538